CLINICAL TRIAL: NCT04128657
Title: Validation of the Morocan Arabic Version of the Low Anterior Resection Syndrome (LARS) Score for Measuring Bowel Dysfunction and Wexner Score of Incontinence After Sphincter-preserving Surgery Among Rectal Cancer Patients
Brief Title: Validation of the Moroccan Arabic Version of the Low Anterior Resection Syndrome (LARS) and Wexner Score of Continence Among Rectal Cancer Patients
Acronym: MA_LARSWEX
Status: Completed | Type: Observational
Sponsor: Moroccan Society of Surgery (Other)
Collaborators: Institut National d'Oncologie Sidi Mohammed Ben Abdellah (Unknown)
Responsible Party: Principal Investigator, Amine Souadka, professor, Moroccan Society of Surgery
Other Study IDs: LARS_Wexner_MA
Record Dates: First submitted 2019-10-13; First posted 2019-10-16 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Rectal Cancer Patients
Keywords: Quality of life; Sphincter sparing surgery; Wexner score; LARS score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MA_LARS — Validation of the MA_LARS and MA_Wexner
  Other Names: MA_Wexner

SUMMARY:
In the past decade, colorectal cancer management improved considerably with total mesorectal excision as well as the multidisciplinary management relying on neoadjuvant radiochemotherapy. This forward leap is currently responsible for an increase in the survivorship of colorectal cancer patients to more than 50% at 5 years. Additively the surgical approach is now more inclined towards sphincter preserving procedures, which allows the conservation of body image but can have negative bowel function repercussions consisting of urgency and incontinence ; all these terms encompassed in the low anterior resection syndrome.

In the light of these findings many studies developed assessment tools in order to objectively measure this functional alteration among which are the low anterior resection syndrome questionnaire (LARS) and the WEXNER score. These tools designed to assess bowel function after sphincter-preserving surgery are now translated and validated into various languages and used in different countries.

The LARS score relies on the frequency of the symptoms and allows the categorization of patients into 3 groups: no LARS (0-20 points), minor LARS (21-29 points), and major LARS (30-42 points). It assesses the frequency of emptying, incontinence ( liquid, gas ), and other symptoms such as urgency and incomplete voiding. On the other hand, the WEXNER score relies on the examination of the frequency of three types of fecal incontinence (solid, liquid, and gas) and their consequences (pad wearing and lifestyle alteration) with frequency options ranging from never (score 0) through to always (meaning at least once per day; score 4). The score ranges from 0 (perfect continence) to 20 (complete incontinence).

The aim of our study is to adapt and validate the LARS and WEXNER score to the moroccan arabic dialect.

DETAILED DESCRIPTION:
The translation of the LARS and WEXNER score to the moroccan dialect ( arabic ) has been done in another study using translation and back translation in concordance with the international guidelines. The questionnaire is administered to a total of 102 patients either directly or via telephone. Reproducibility will be tested through test and retest as one sub-group will be administered the questionnaire twice with an interval of 1 to 2 weeks. Patients will also be administered the questionnaires of the European Organization for Research and treatment of Cancer (EORTC) : QLQ-C30.

The validity of the LARS and WEXNER score will be tested by using the indicators of discriminant validity and convergent validity which will be determined in this study by computing the correlations between the LARS and WEXNER scores to the EORTC QLQ-C30.

For discriminant validity testing, variables used will be factors known to affect bowel function after colorectal surgery such as gender, age, neoadjuvant therapy, distance of the tumor from the anal verge, prior temporary stoma, length of postoperative period, the need for a reintervention and the occurrence of complications.

We recruited for our study patients treated in the National Oncology Institute of Rabat and in the Al azhar oncology center in the surgical department of Pr. Souadka Abdelilah with a minimum post operative interval of 6 months.

The validation of a moroccan dialectical version of the LARS score and WEXNER score will allow a better understanding of the bowel function post surgery and thereby the identification of patients with the highest scores which will allow a better understanding and possible inclusion of these tools in patient outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged older than 18 years.
* Neoplasm of the rectum.
* Rectal cancer patients undergoing curative sphincter-preserving surgery with (partial or total) mesorectal excision.
* Surgery performed between January 2012 to March 2019, with reversal of the defunctioning stoma before March 2019;
* Bowel continuity restoration for at least 6 months.
* Consent to participate in the study.

Exclusion Criteria:

* Palliative surgery.
* The presence of a definitive iliac or perineal stoma.
* Diseases of bowel dysfunction (Crohn's disease)
* Cognitive and/or language issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volantary patient with curative sphincter preserving surgery with no defuntioning stoma who accept to participate in the MA_LARS and MA_Wexner scores validation study
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Validation of the moroccan arabic version of the LARS score | 6 months after surgery
  Validation of the Moroccan arabic Low anterior resection syndrome (LARS) score ; 0 to 20 (no LARS), 21 to 29 (minor LARS ) and 30 to 42 (Major LARS )
Validation of the moroccan arabic version of the Wexner score | 6 months after surgery
  validation of the Moroccan arabic Wexner score; 0 perfect score and 20 complete incontinence

CONTACTS AND LOCATIONS:
Locations (2):
- Morocco (2):
  - National Institut of Oncology, Surgical oncology department, Rabat, Please Enter the State Or Province
  - Private surgical oncology center, Salé

IPD SHARING:
Plan to Share IPD: Undecided